CLINICAL TRIAL: NCT02723526
Title: Development of a Prognostic Model for Metastatic Hormone-sensitive Prostate Cancer by Sequentially Analyzing the Expression of Tumor Markers in Circulating Tumor Cells
Brief Title: Expression of Tumor Markers in Circulating Tumor Cells of Metastatic Hormone-sensitive Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Bo Dai, Clinical Professor of Department of Urology, Fudan University
Other Study IDs: CTC-mHSPC
Record Dates: First submitted 2016-03-26; First posted 2016-03-30 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Prostate Cancer
Keywords: Metastatic Hormone-Sensitive Prostate Cancer；circulating tumor cells；Prognosis；Liquid biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single arm
  Interventions: Other: Blood drawing

INTERVENTIONS:
Other: Blood drawing

SUMMARY:
As prostate cancer progresses, tumor cells dissociate and enter the bloodstream. Considered a "liquid biopsy," these circulating tumor cells (CTC) can show how a patient's cancer evolves and responds to treatments. The purpose of this study is to determine whether sequentially analyzing the expression of tumor markers in circulating tumor cells in newly diagnosed metastatic hormone-sensitive prostate cancer patients can predict the outcome of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients;
2. 18 yrs and older, and 80 yrs and younger;
3. Histologically or cytologically proven prostate adenocarcinoma;
4. Imaging examinations including Emission Computed Tomography (ECT),Positron Emission Tomography (PET),Computed Tomography(CT)and Magnetic Resonance Imaging (MRI) revealed non-regional lymph node metastasis, bone metastasis, or visceral metastasis;
5. Not yet receiving hormonal therapy;
6. Not yet receiving chemotherapy previously;
7. Not yet receiving radical prostatectomy, radiotherapy, or transurethral resection of the prostate (TURP) previously;
8. Patients are willing to participate and can be followed up regularly；

Exclusion Criteria:

1. Received radical prostatectomy, radiotherapy, or transurethral resection of the prostate (TURP) previously;
2. Received androgen deprivation therapy (including surgical castration, medical castration, anti-androgen therapy, and maximum androgen blockade) before inclusion;
3. Patients received chemotherapy previously;
4. Combined with other malignant tumor history (in addition to the skin basal cell carcinoma or other tumors that have been cured more than five years);

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly Diagnosed Metastatic Hormone-Sensitive Prostate Cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
time to castration-resistant prostate cancer | 3 years

SECONDARY OUTCOMES:
time to radiographic progression | 3 years
time to prostate specific antigen (PSA) progression | 3 years
time to prostate specific antigen (PSA) nadir | 2 years
complete serologic response rate at 6 month and 12 month | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Bo Dai, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No